CLINICAL TRIAL: NCT06629090
Title: Cerebrovascular Responses to Acute Hypoperfusion
Brief Title: Brain Blood Vessel Responses to Changes in Blood Flow: Younger Cohort
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-0377: Younger Cohort; A176000 (Other: UW- Madison); EDUC/KINESIOLOGY (Other: UW- Madison); Protocol Version 7/29/2025 (Other: UW- Madison)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Magnetic Resonance Imaging; Cerebrovascular Circulation
Keywords: Magnetic Resonance Imaging; Brain Blood Flow; Lower Body Negative Pressure; Carbon Dioxide
MeSH Terms: interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Young Adults (Experimental): Young Adults between 20-40 years of age.
  Interventions: Device: MRI; Drug: Prazosin; Drug: Placebo

INTERVENTIONS:
Device: MRI — Participants will undergo an MRI scan while performing breathing and simulated postural change tasks.
Drug: Prazosin — A dose of prazosin will be administered based on body weight
Drug: Placebo — Oral placebo

SUMMARY:
Brain blood flow will be measured during a simulated postural change test and while breathing increased levels of carbon dioxide using magnetic resonance imaging.

DETAILED DESCRIPTION:
Global cerebral blood flow (CBF) decreases with advancing age; however, some adults have accelerated declines in CBF, placing them at a greater risk of cognitive impairment. However, there is a lack of human studies that investigate the cause or consequence of altered blood flow regulation in the brain. This study will systematically address this gap in knowledge by examining cerebrovascular control in adults during acute physiological challenges (simulated postural change test and breathing increased carbon dioxide) that stimulate a change in CBF.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-40 years
* Have a BMI ≤34.5 kg/m2
* are less than 72 in (182.88 cm) height
* Nonsmoker

Exclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (MCI) or Alzheimer's disease (AD)
* History or evidence of hepatic disease, hematological disease, or peripheral vascular disease; severe kidney injury requiring hemodialysis
* History of cardiovascular disease including: severe congestive heart failure, coronary artery disease, ischemic heart disease (stents, coronary artery bypass grafts) and tachycardia
* Uncontrolled hypertension
* History of clinically significant ischemic or hemorrhagic stroke, or significant cerebrovascular disease
* Severe untreated obstructive sleep apnea
* History of diabetes with HbA1c greater than 9.5 percent
* Major neurologic disorders other than dementia (e.g., MS, ALS, brain surgery, etc.)
* Current or recent (less than1 year) major psychiatric condition (Axis I) or addictive disorders
* Significant surgical history
* Other significant medical conditions at investigators' discretion
* Contraindications to MRI
* Prescribed medications that interfere with prazosin
* Lactose allergy
* lower body will not fit in lower body negative pressure (LBNP) chamber (regardless of overall height and BMI)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood velocity | Two study visits, up to 240 minutes
  The change in blood velocity during breathing and simulated postural change tasks will be measured with MRI
Change in blood flow | Two study visits, up to 240 minutes
  The change in intracranial blood flow during breathing and simulated postural change tasks will be measured with MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jill Barnes, PhD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No